CLINICAL TRIAL: NCT01237171
Title: Outcome Study of Cesium-131 Brachytherapy Following Sub-Lobar Resection for Early Stage NSCLC
Brief Title: A Study of Cesium-131 Brachytherapy Following Sub-Lobar Resection for Early Stage Non Small Cell Lung Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Study never moved past ideation phase
Sponsor: IsoRay Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Cs131-Lung001
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: NSCLC; Non Small Cell Lung Cancer
Keywords: Brachytherapy; Lung Brachytherapy; NSCLC; Sub-lobar resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sub-lobar resection with Cesium-131: All enrolled patients will undergo sub-lobar resection and brachytherapy implant with Cesium-131 in an effort to study and quantify recurrence/control patterns.
  Interventions: Radiation: Cesium-131 Brachytherapy Seed

INTERVENTIONS:
Radiation: Cesium-131 Brachytherapy Seed — 85 Gray Dose
  Other Names: Sealed Brachytherapy Source CS-1 (IsoRay Medical)

SUMMARY:
For patients diagnosed with early (Stage I) non-small cell lung cancer, a lobe of lung is usually removed at surgery to treat the cancer. For some patients, the removal of a lobe of lung may leave too little lung behind for easy breathing. For some of these patients, it may be possible to perform a smaller-scale surgery ("sub-lobar resection") and place a radioactive implant behind to prevent the cancer from growing back. This study will see how these patients do in terms of controlling their disease treated with a radioactive implant called Cesium-131.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have suspicious lung nodule for clinical stage I/recurrent non-small cell Lung Cancer
2. Mass Tumor size < 7 cm
3. Patient must have a CT scan of the chest with upper abdomen within 90 days prior to date of pre-registration.
4. Patient must have ECOG/Zubrod performance status 0,1, or 2.

Exclusion Criteria:

1. Patient has already received high dose radiation to the area
2. Cancerous nodule is very close to the esophagus or spinal cord, thereby increasing the risk of radiation treatment
3. Pregnancy or unwillingness to practice a form of birth control (i.e. abstinence, oral contraceptives, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinical stage I non-small cell lung cancer who are not candidates for full lobectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11 (Estimated); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Local Recurrence | 3 Years
  Cancer regrowth in the area where it was surgically removed

SECONDARY OUTCOMES:
Quality of Life | 2 years
  Using questionnaires, data will be collected related to the sense of well-being experienced by the patient after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bhupesh Parashar, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States